CLINICAL TRIAL: NCT00250718
Title: Phase II Study: Treatment of Relapsed Lymphoid Malignancies With an Anti-angiogenic Approach
Brief Title: Study: Treatment of Relapsed Lymphoid Malignancies With an Anti-Angiogenic Approach
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low rate of accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1003C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Non-Hodgkin's Lymphoma; Cancer
Keywords: Non Hodgkin's Lymphoma; Phase II; Lymphoid malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — Vincristine; Etoposide; Rituximab; Dexamethasone; Calcium Dobesilate; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 Combination Treatment (Experimental): Treatment with combination therapy as follows:
  VP-16 at 50 mg/day, orally for 14 days every 28 days; Chlorambucil at 0.1 mg/kg/day orally for 14 days every 28 days; Vincristine at 2 mg intravenously every 14 days; Dexamethasone at 200 mg intravenously every 24 days; Rituxan (rituximab) at 375 mg/m2 intravenously every 14 day; Levofloxacin at 500 mg orally daily; Diflucan at 200 mg orally daily
  At least 2 courses, but no more than 8 courses total, will be administered to each patient
  Interventions: Drug: Vincristine; Drug: VP-16; Drug: Rituximab; Drug: Dexamethasone; Drug: Levofloxacin

INTERVENTIONS:
Drug: Vincristine — Vincristine should be administered intravenously through a freely-running IV.
  Other Names: Oncovin
Drug: VP-16 — The VP-16 is optional for the first cycle if the patient has delays in obtaining the drug.
  Other Names: Etoposide; NSC-67574; Vepesid; Ethylidene-Lignan P
Drug: Rituximab — The total amount of rituximab needed for a patient's entire infusions (one course) will be determined at study entry. A single dose of 375 mg/m2 will be based upon the patient's actual body surface area calculated during the baseline evaluation. The dose level of rituximab will not be adjusted.
  Patients will only receive rituximab if their tumors are CD20 positive CLL or NHL.
  Rituximab will only be administered to patients if they have previously had less than 8 doses. If a patient is treated with rituxan they should have at least 4 doses
  Other Names: Rituxan
Drug: Dexamethasone — Dexamethasone will be administered at 200mg q 14 days. Dexamethasone should be administered over a 1 hour infusion.
  Other Names: decadron
Drug: Levofloxacin — Levofloxacin will be administered at 500 mg PO qd.
  Other Names: Levaquin; Levaquin Leva-Pak

SUMMARY:
1.1 To determine the efficacy of a combination treatment of VP-16, chlorambucil, dexamethasone, and vincristine in patients with relapsed/refractory hematological malignancies.

1.2 To determine the toxicity profile of the above regimen in this patient population.

1.3 Evaluate the effect of low dose administration of chemotherapy on angiogenesis, and correlate this with tumor responses.

DETAILED DESCRIPTION:
The purpose of the study is to see how effective the combination of chemotherapy drugs VP-16, chlorambucil, dexamethasone, and vincristine is for patients who have blood cancers that have returned or not responded to prior treatment. Some patients may also receive a medication called rituximab if their doctor thinks it is appropriate. This drug combination will be given to study participants in a low dose continuous basis. The study will also collect information about the side effects of the above drug combination on patients with these types of cancers. Previous studies on patients with non-Hodgkin's lymphoma indicate that some patients treated with this drug combination achieved a high response. The aim of this study is to test this drug combination in a controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, with Hodgkin's lymphoma, Non-Hodgkin lymphoma (NHL), multiple myeloma (MM), or chronic lymphocytic leukemia (CLL) are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,000 or cells/mm3 and platelet count >50,000/mm3 and absence of a regular red blood cell or platelet transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 2.0 x upper limit of normal.
* Patients must have received at least two previous chemotherapy regimens for their disease.
* Patients must have measurable disease (NHL) or evaluable disease (MM, CLL).

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dulcinea Quintana, MD, Principal Investigator — UNM Cancer Center; Robert Hromas, MD, Study Chair — University of Florida
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: UNM Cancer Center — http://www.cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Combination Treatment: VP-16 at 50 mg/day, orally for 14 days every 28 days; Chlorambucil at 0.1 mg/kg/day orally for 14 days every 28 days; Vincristine at 2 mg intravenously every 14 days; Dexamethasone at 200 mg intravenously every 24 days; Rituxan (rituximab) at 375 mg/m2 intravenously every 14 day; Levofloxacin at 500 mg orally daily; Diflucan at 200 mg orally daily
  One cycle lasts 28 days. At least 2 but no more than 8 cycles will be administered to each patient
Period: Overall Study
Arm/Group | Arm 1 Combination Treatment
Started | 17
Received Treatment | 16
Completed | 14
Not Completed | 3
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 Combination Treatment
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Sum of Complete and Partial Responses
Description: Solid tumor response is per Response Evaluation Criteria in Solid Tumors (RECIST) (ver 1.0).
  For CLL: complete remission (CR) requires the following for>=2 months 1) no symptoms attributable to CLL, 2) normal physical examination, 3) absolute lymphocyte count<4,000/µL, 4) ANC>1,500/µL, 5) platelets>100,000/µL, 6) hemoglobin>11 g/dL, 7) bone marrow lymphocytosis<30%, 8) no nodules in bone marrow. Partial response (PR) requires the following for >=2 months 1) decrease in previously enlarged nodes, spleen, and liver by >=50%, 2) ANC>=1,500/µL or platelets>=100,000/µL, 3) hemoglobin>=11 g/dL, 4) 50% improvement over pre-therapy reductions in hemoglobin and/or platelets.
  For MM, CR is no monoclonal protein (M-protein) in blood and urine and <5% plasma cells in bone marrow on >=2 determinations >=6 wk apart & stable bone disease & calcium levels. PR is>50% and >90% decreases in serum & urine M-protein, respectively, on >=2 occasions for >=6 wk, stable bone disease & calcium.
Time Frame: Up to 6 months after first on-study treatment
Population: Trial was terminated due to low accrual; no data to report. An insufficient number of subjects were accrued to report data accurately.
Arm/Group | Arm 1 Combination Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity
Time Frame: End of 2 cycles (cycle = 28 days)
Population: Trial was terminated early due to low accrual; no data to report. Adverse event data for enrolled patients is reported in the adverse event results section.
Arm/Group | Arm 1 Combination Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Arm 1 Combination Treatment: VP-16 50mg/d PO x14 days q 28 days + Chlorambucil 0.1mg/kg/d PO x14 days q 28 days + Vincristine 2mg IV x14 days + Dexamethasone 200mg IV q 24 days + Rituxan (rituximab) 375 mg/m2 IVI x14 days + Levofloxacin 500 mg PO qd + Diflucan 200 mg PO qd
  Vincristine: should be administered intravenously through a freely-running IV at 2mg q 14 days.
  VP-16: The VP-16 is optional for the first cycle if the patient has delays in obtaining the drug. Dose and schedule 50 mg/d P.O. x14 days q 28 days.
  Rituximab: The total amount of rituximab needed for a patient's entire infusions (one course) will be determined at study entry. A single dose of 375 mg/m2 will be based upon the patient's actual body surface area calculated during the baseline evaluation. The dose level of rituximab will not be adjusted.
  Dexamethasone: Dexamethasone will be administered at 200mg q 14 days. Dexamethasone should be administered over a 1 hour infusion.
  Levofloxacin: Levofloxacin will be administ
Arm/Group | Arm 1 Combination Treatment
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Combination Treatment (N=16)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (2)
Arrhythmia (irregular heartbeat) (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Hyperglycemia (high blood sugar) (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Combination Treatment (N=16)
Allergic rhinitis (runny nose) (Immune system disorders) | 1 (1)
Tinnitus (ringing in the ears) (Ear and labyrinth disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (20)
Leukocytes decreased (Blood and lymphatic system disorders) | 5 (23)
Neutrophils decreased (Blood and lymphatic system disorders) | 7 (28)
Platelet count decreased (Blood and lymphatic system disorders) | 5 (10)
Hypotension (low blood pressure) (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 11 (14)
Fever (General disorders) | 3 (3)
Rigors (stiffness) (General disorders) | 1 (1)
Increased sweating (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 4 (4)
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Taste disturbance (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Epistaxis (Nosebleed) (General disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Edema: limbs (General disorders) | 1 (1)
Hypercalcemia (High calcium levels) (Investigations) | 1 (2)
Hyperglycemia (High blood glucose) (Investigations) | 2 (3)
Hyperuricemia (High uric acid) (Investigations) | 1 (3)
Hypoalbuminemia (Low albumin levels) (Investigations) | 1 (1)
Hypocalcemia (Low calcium levels) (Investigations) | 1 (1)
Hypokalemia (Low potassium levels) (Investigations) | 5 (6)
Hypomagnesemia (Low magnesium levels) (Investigations) | 1 (4)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Agitation (Nervous system disorders) | 2 (3)
Anxiety (Nervous system disorders) | 2 (3)
Ataxia (Lack of muscle coordination) (Nervous system disorders) | 1 (1)
Confusional state (Nervous system disorders) | 2 (2)
Convulsions (Nervous system disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 3 (3)
Neurology - Other (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Extraocular muscle disorder (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (3)
Abdominal pain (General disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Chest pain (General disorders) | 1 (1)
Myalgia (Muscle pain) (Musculoskeletal and connective tissue disorders) | 3 (3)
Neuralgia (Nerve pain) (Nervous system disorders) | 1 (17)
Pain - Other (General disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (10)
Scrotal pain (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Decreased libido (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No